CLINICAL TRIAL: NCT01422772
Title: Open-label, Non-comparative, Dose-escalation, Single-center, Phase 1 Trial to Evaluate the Safety of VM202RY Gene Medicine Injected Into Cardiac Muscle of Incompletely Revascularized Area After CABG in Patients With Ischemic Heart Diseases
Brief Title: Safety Study of Gene Therapy for Ischemic Heart Disease in Korea
Acronym: Engensis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VM202RY-VM01
Record Dates: First submitted 2011-08-21; First posted 2011-08-24 (Estimated); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Heart Disease
Keywords: VM202; Engensis; Coronary Artery Bypass Graft
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: Dose-escalation
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort I (Experimental): 0.5 mg/ 1 mL of VM202 was intramyocardially injected into 4 sites
  Interventions: Biological: VM202-0.5 mg
- Cohort II (Experimental): 1 mg/ 2 mL of VM202 was intramyocardially injected into 8 sites
  Interventions: Biological: VM202-1.0 mg
- Cohort III (Experimental): 2 mg/ 4 mL of VM202 was intramyocardially injected into 8 sites
  Interventions: Biological: VM202-2.0 mg

INTERVENTIONS:
Biological: VM202-0.5 mg — 0.5 mg intramyocardial injection
  Arms: Cohort I
Biological: VM202-1.0 mg — 1 mg intramyocardial injection
  Arms: Cohort II
Biological: VM202-2.0 mg — 2 mg intramyocardial injection
  Arms: Cohort III

SUMMARY:
The purpose of this study is to evaluate the safety of VM202 (Engensis) direct injection into the cardiac muscles of the coronary artery territory where complete revascularization could not be done even through Coronary Artery Bypass Graft (CABG).

DETAILED DESCRIPTION:
All the patients expected to undergo Coronary Artery Bypass Graft (CABG) will screen for the participation in the clinical study. Subjects who signed the informed consent will receive all the screening tests within 21 days before surgery (Day 0). VM202 (Engensis) will be injected into 4 sites or 8 sites on the coronary artery where complete revascularization was not done since vascular anastomosis could not be performed due to the bad vascular condition during surgery. VM202 (Engensis) will be administered to Group1 (0.5 mg), Group 2 (1 mg) and Group 3 (2 mg) at different concentrations. Subjects will be scheduled to get inpatient treatment during the gene therapy period (7 days) and follow-up tests at Week 2, 4, 8, 12 and 24 based on surgery day (Day 0). Adverse events and concomitant drugs will be checked.

Safety: Evaluated for 6 months after the administration of VM202 (Engensis).

1. Dose-Limiting Toxicity (DLT)
2. Tolerated Dose (TD)
3. Adverse events, vital signs, physical examination and laboratory test values
4. Major Adverse Cardiac Event (MACE) - cardiac death, myocardial infarction, ventricular arrhythmia requiring treatment, or hospitalization for revascularization of target blood vessels)
5. Safety of VM202 intramyocardial injection: persistent hemorrhage, arrhythmia and other complications

Secondary endpoints

- Efficacy

1. Changes in cardiac function: Left ventricular ejection fraction and cardiac function in the local region by cardiac MRI (Magnetic Resonance Imaging), myocardial SPECT (99 mTc Sestamibi Methoxyl Isobutyl Isonitrile Single Photon Emission Computed Tomography) and Trans Thoracic echocardiography (TTE)
2. Size of viable myocardium: By cardiac MRI (myocardial thickness of intramyocardial gene injection site, gadolinium late contrast enhancement range and the exercise intensity of the local region)
3. Changes in myocardial ischemic area: By myocardial SPECT (blood flow changes at intramyocardial gene injection site from resting to stress condition)

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 19 and ≤ 75 years
2. Patients in whom decrease of myocardial perfusion in coronary artery territories (rest perfusion - stress perfusion: ≥ 7%) was observed by myocardial SPECT
3. Patients judged to have possibly incomplete revascularization based on the observation of the coronary artery's internal diameter of ≤ 1 mm, diffuse atherosclerosis or severe calcification on coronary angiography, or patients judged to have some myocardial perfusion territories that could not be performed Coronary Artery Bypass Graft
4. Patients who or whose legal representative can write the informed consent before the initiation of the clinical study and comply with the requirements

Exclusion Criteria:

1. Patients with progressive or present heart failure
2. Patients with uncontrolled ventricular arrhythmia on electrocardiogram, or who have been treated for ventricular arrhythmia
3. Patients with current or history of malignant tumor
4. Patients with severe infectious disease
5. Patients with uncontrolled hematologic disorders
6. Patients requiring surgery for the accompanying valve diseases or left ventricular volume reduction surgery
7. Patients with current or history of proliferative retinopathy
8. Patients with remaining life of less than 1 year and severe accompanying diseases enough to die during the clinical follow-up period
9. Patients with history of drug or alcohol abuse within the recent 3 months
10. Women who are pregnant or breast feeding or postmenopausal women of childbearing age. However, women who underwent surgical sterilization including hysterectomy or bilateral tubal ligation can participate in this clinical trial. Even though they consent to the contraception, they cannot be enrolled.
11. Patients in inappropriate condition judged by investigators
12. Patients with cerebrovascular diseases (cerebral infarction, cerebral bleeding or transient ischemic attack that are currently occurring or occurred within 6 months)
13. Patients with idiopathic hypertension who are not controlled with drugs
14. Patients with severe hepatic disorders
15. Patients with severe renal disorders
16. Patients who underwent Coronary Artery Bypass Graft
17. Patients who underwent angioplasty within 1 year before their enrollment in the study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gibong Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Kim JS, Hwang HY, Cho KR, Park EA, Lee W, Paeng JC, Lee DS, Kim HK, Sohn DW, Kim KB. Intramyocardial transfer of hepatocyte growth factor as an adjunct to CABG: phase I clinical study. Gene Ther. 2013 Jul;20(7):717-22. doi: 10.1038/gt.2012.87. Epub 2012 Nov 15. PMID 23151518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 participants were screened. 9 participants were randomized/enrolled, with 7 screen failures.
Groups:
- Group 1 - 0.5 mg/1 mL: VM202 (Engensis) 0.5 mg/1 mL was intramyocardially injected into 4 sites 0.125 mg/0.25 mL/injection point) of the incompletely revascularized area after Coronary Artery Bypass Graft.
- Group 2 - 1.0 mg/2 mL: VM202 (Engensis) 1 mg/2 mL was intramyocardially injected into 8 sites (0.125 mg/0.25 mL/injection point) of the incompletely revascularized area after Coronary Artery Bypass Graft.
- Group 3 - 2 mg/4 mL: VM202 (Engensis) 2 mg/4 mL was intramyocardially injected into 8 sites (0.25 mg/0.5 mL/injection point) of the incompletely revascularized area after Coronary Artery Bypass Graft.
Period: Overall Study
Arm/Group | Group 1 - 0.5 mg/1 mL | Group 2 - 1.0 mg/2 mL | Group 3 - 2 mg/4 mL
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat
Groups:
- Group 1 - VM202 - 0.5 mg/ 1mL: VM202RY 0.5 mg/ 1 mL was intramyocardially injected into 4 sites (0.125 mg/0.25 mL/injection point) of the incompletely revascularized area after Coronary Artery Bypass Graft.
- Group 2 - VM202 - 1.0 mg/2 mL: VM202RY 1 mg/2 mL was intramyocardially injected into 8 sites (0.125 mg/0.25 mL/injection point) of the incompletely revascularized area after Coronary Artery Bypass Graft.
- Group 3 - VM202 - 2 mg/4 mL: VM202RY 2 mg/4 mL was intramyocardially injected into 8 sites (0.25 mg/0.5 mL/injection point) of the incompletely revascularized area after Coronary Artery Bypass Graft.
- Total: Total of all reporting groups
Arm/Group | Group 1 - VM202 - 0.5 mg/ 1mL | Group 2 - VM202 - 1.0 mg/2 mL | Group 3 - VM202 - 2 mg/4 mL | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.00 (12.77) | 59.00 (6.93) | 67.67 (6.11) | 62.56 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3
  Male | 2 | 3 | 1 | 6
Region of Enrollment [Number; unit: participants]
  South Korea | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Adverse Events - Total Adverse Events (AE)
Description: Subjects who have been administered the investigational drug will be included, regardless of protocol violations or adherence to visit schedules. This clinical trial is designed to evaluate safety over a 6-month period.
  Assessments Include:
  Adverse reactions, vital signs, physical exam, laboratory test results
Time Frame: 24 weeks
Population: Total Number of Adverse Events (ITT Safety)
Measure: Number; unit: Total AEs
Units Other Than Participants: Total AEs
Arm/Group | Group 1 - 0.5 mg/1 mL | Group 2 - 1.0 mg/2 mL | Group 3 - 2 mg/4 mL
Number analyzed (Participants) | 3 | 3 | 3
Number analyzed (Total AEs) | 60 | 18 | 36
Total AEs
  Treatment Emergent AEs | 58 | 18 | 36
  AEs related to Investigational Product | 0 | 0 | 0
  Serious Adverse Events | 2 | 0 | 0

2. Primary Outcome: The Severity of Adverse Events - Total Adverse Events by Severity
Description: as for outcome 1
Time Frame: 24 weeks
Population: Total Adverse Events by Severity (ITT Safety)
Measure: Number; unit: Total AEs
Arm/Group | Group 1 - 0.5 mg/1 mL | Group 2 - 1.0 mg/2 mL | Group 3 - 2 mg/4 mL
Number analyzed (Participants) | 3 | 3 | 3
Total AEs
  Grade 1/Mild-Severity of AEs | 31 | 6 | 12
  Grade 2/Moderate-Severity of AEs | 27 | 12 | 24
  Grade 3/Severe-Severity of AEs | 0 | 0 | 0
  Grade 4/Severe-Severity of AEs | 0 | 0 | 0

3. Secondary Outcome: Percentage of Change From Baseline/Screening in Left Ventricular Ejection Fraction Evaluated by Magnetic Resonance Imaging
Description: Changes in Percentage of Left Ventricular Ejection Fraction by Cardiac Magnetic Resonance Imaging (MRI). Cardiac MRI will be used to monitor for the development of intramyocardial hemangiomas. Analysis will follow the standard cardiac MRI protocols of the Department of Radiology at Seoul National University Hospital, using an appropriate segment model based on the patient's heart size. Parameters evaluated will include left ventricular volume (mL), wall motion index, myocardial thickness (mm), and LVEF (%). Comparisons will be made between baseline/screening and follow-up measurements for each patient, as well as between treatment groups.
Time Frame: Day 0, 12 weeks, 24 weeks
Population: Intent to Treat - Left Ventricular Ejection Percentage Fraction - Measured by Magnetic Resonance Imaging (MRI)
Measure: Mean (Standard Deviation); unit: percentage of change from screening
Arm/Group | Group 1 - 0.5 mg/1 mL | Group 2 - 1.0 mg/2 mL | Group 3 - 2 mg/4 mL
Number analyzed (Participants) | 3 | 3 | 3
percentage of change from screening
  Week 12 | 1.77 (6.54) | 1.63 (6.96) | 2.67 (5.12)
  Week 24 | 0.45 (3.89) | 6.80 (6.93) | 0.13 (11.19)

4. Secondary Outcome: Percentage of Change From Baseline/Screening in Cardiac Function Evaluated by Echocardiography
Description: Changes from screening in cardiac function evaluated based on Percentage of Left Ventricular Ejection Fraction by cardiac Trans-thoracic Echocardiography (TTE). From transthoracic echocardiography, left ventricular diameter (mm), ejection fraction (%), and wall thickness (mL) will be measured and compared from Screening/Baseline to follow-up results after surgery. The Wall Motion Score Index will be calculated by dividing the myocardium into 16 segments and assigning a score to each area based on motion: [1 = normal, 2 = hypokinetic, 3 = akinetic, 4 = dyskinetic]. The total score for the entire myocardium and the right coronary artery region will be averaged by the number of segments.
Time Frame: Day 0, Day 7, 12 weeks, 24 weeks
Population: Intent to Treat - Left Ventricular Ejection Percentage Fraction - Measured by Trans Thoracic Echocardiography
Measure: Mean (Standard Deviation); unit: percentage of change from screening
Arm/Group | Group 1 - 0.5 mg/1 mL | Group 2 - 1.0 mg/2 mL | Group 3 - 2 mg/4 mL
Number analyzed (Participants) | 3 | 3 | 3
percentage of change from screening
  Day 7 | -1.00 (2.65) | 0.0 (2.0) | -1.0 (3.0)
  Week 12 | 3.0 (6.08) | -2.0 (4.58) | -1.33 (3.79)
  Week 24 | 8.0 (4.24) | 3.0 (12.12) | 3.33 (11.93)

5. Secondary Outcome: Changes in Size of Viable Myocardium - End-Systolic Thickness
Description: The size of the viable myocardium was evaluated based on the myocardium thickness at the site of intramyocardial gene injection by Magnetic Resonance Imaging - End-Systolic Thickness. Using cardiac MRI, the myocardial thickness at the gene injection site, the extent of late gadolinium enhancement, and local wall motion strength will be evaluated. Differences between groups before and after VM202RY administration will be tested using the Kruskal-Wallis test.
Time Frame: Day 0, 12 weeks, 24 weeks
Population: Intent to Treat - myocardium thickness by Magnetic Resonance Imaging - End-Systolic Thickness
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group 1 - 0.5 mg/1 mL | Group 2 - 1.0 mg/2 mL | Group 3 - 2 mg/4 mL
Number analyzed (Participants) | 3 | 3 | 3
mm
  Week 12 | 0.58 (1.40) | 0.08 (1.67) | 0.93 (1.37)
  Week 24 | 0.99 (2.59) | 0.36 (1.63) | 1.15 (1.38)

6. Secondary Outcome: Changes in Size of Viable Myocardium - End-Diastolic Thickness
Description: The size of the viable myocardium was evaluated based on the myocardium thickness at the site of intramyocardial gene injection by Magnetic Resonance Imaging - End-Diastolic Thickness. Using cardiac MRI, the myocardial thickness at the gene injection site, the extent of late gadolinium enhancement, and local wall motion strength will be evaluated. Differences between groups before and after VM202RY administration will be tested using the Kruskal-Wallis test.
Time Frame: Day 0, 12 weeks, 24 weeks
Population: Intent to Treat - myocardium thickness by Magnetic Resonance Imaging - End-Diastolic Thickness
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group 1 - 0.5 mg/1 mL | Group 2 - 1.0 mg/2 mL | Group 3 - 2 mg/4 mL
Number analyzed (Participants) | 3 | 3 | 3
mm
  Week 12 | 0.47 (1.13) | 0.71 (0.23) | 0.44 (0.46)
  Week 24 | 1.85 (0.10) | 0.43 (1.53) | 0.17 (0.81)

7. Secondary Outcome: Changes in Myocardial Ischemic Area - Stress Condition
Description: Changes in Myocardial Ischemic Area evaluated by 99mTc Sestamibi Methoxyl Isobutyl Isonitrile Single Photon Emission Computed Tomography (SPECT) based on Percentage of perfusion volume - Stress Condition
Time Frame: Day 0, 12 weeks, 24 weeks
Population: Intent to Treat - Changes in Myocardial Ischemic Area evaluated by SPECT based on Percentage of perfusion volume - Stress Condition
Measure: Mean (Standard Deviation); unit: percentage of Perfusion Volume
Arm/Group | Group 1 - 0.5 mg/1 mL | Group 2 - 1.0 mg/2 mL | Group 3 - 2 mg/4 mL
Number analyzed (Participants) | 3 | 3 | 3
percentage of Perfusion Volume
  Week 12 | 7.83 (7.91) | 8.33 (1.53) | 1.67 (7.75)
  Week 24 | 7.50 (7.07) | 5.00 (1.50) | 5.33 (8.13)

8. Secondary Outcome: Changes in Myocardial Ischemic Area - Resting Condition
Description: Changes in Myocardial Ischemic Area evaluated by 99mTc Sestamibi Methoxyl Isobutyl Isonitrile Single Photon Emission Computed Tomography (SPECT) based on Percentage of perfusion volume - Resting Condition
Time Frame: Day 0, 12 weeks, 24 weeks
Population: Intent to Treat - Changes in Myocardial Ischemic Area evaluated by SPECT based on Percentage of perfusion volume - Resting Condition
Measure: Mean (Standard Deviation); unit: percentage of Perfusion Volume
Arm/Group | Group 1 - 0.5 mg/1 mL | Group 2 - 1.0 mg/2 mL | Group 3 - 2 mg/4 mL
Number analyzed (Participants) | 3 | 3 | 3
percentage of Perfusion Volume
  Week 12 | 7.33 (8.50) | 0.83 (1.53) | 4.67 (4.86)
  Week 24 | -3.50 (0.71) | 1.33 (2.75) | 5.17 (10.41)

ADVERSE EVENTS:
Time Frame: 6 months
Description: The incidence and the number of cases for all the treatment-emergent AEs and the investigational product-related ADRs
Groups:
- Group 1 - VM202 - 0.5 mg/ 1mL: VM202RY 0.5mg/1mL was intramyocardially injected into 4 sites
- Group 2 - VM202 - 1.0 mg/2 mL: VM202RY 1mg/2mL was intramyocardially injected into 8 sites
- Group 3 - VM202 - 2 mg/4 mL: VM202RY 2mg/4mL was intramyocardially injected into 8 sites
Arm/Group | Group 1 - VM202 - 0.5 mg/ 1mL | Group 2 - VM202 - 1.0 mg/2 mL | Group 3 - VM202 - 2 mg/4 mL
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - VM202 - 0.5 mg/ 1mL (N=3) | Group 2 - VM202 - 1.0 mg/2 mL (N=3) | Group 3 - VM202 - 2 mg/4 mL (N=3)
Worsening Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Musculoskeletal and connective tissue disorders spinal column stenosis
Infectious Spondylitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Infections and infestations Infective spondylitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - VM202 - 0.5 mg/ 1mL (N=3) | Group 2 - VM202 - 1.0 mg/2 mL (N=3) | Group 3 - VM202 - 2 mg/4 mL (N=3)
Supraventricular extrasystoles (Cardiac disorders) | 3 (4) | 1 (1) | 2 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 3 (5)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wound Complication (Injury, poisoning and procedural complications) | 1 (3) | 3 (3) | 3 (3)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinopathy hypertensive (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (4) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Periphery motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective spondylitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-01-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT01422772/Prot_SAP_000.pdf